CLINICAL TRIAL: NCT02915744
Title: A Phase 3 Open-Label, Randomized, Multicenter Study of NKTR-102 Versus Treatment of Physician's Choice (TPC) in Patients With Metastatic Breast Cancer Who Have Stable Brain Metastases and Have Been Previously Treated With an Anthracycline, a Taxane, and Capecitabine
Brief Title: A Study of Etirinotecan Pegol (NKTR-102) Versus Treatment of Physician's Choice (TPC) in Patients With Metastatic Breast Cancer Who Have Stable Brain Metastases and Have Been Previously Treated With an Anthracycline, a Taxane, and Capecitabine
Acronym: ATTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-102-14
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Metastasis; Breast Cancer
Keywords: Breast Cancer Brain Metastases (BCBM); Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Carcinoma | interventions — etirinotecan pegol; eribulin; ixabepilone; Vinorelbine; Gemcitabine; Paclitaxel; Docetaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NKTR-102 (Experimental): In Group A, NKTR-102 will be administered at a dose level of 145 mg/m2 on a q21d schedule as a 90-minute intravenous (IV) infusion on Day 1 of each treatment cycle.
  Interventions: Drug: NKTR-102
- Treatment of Physician's Choice (TPC) (Active Comparator): In Group B, TPC will be administered per standard of care. Patients randomized to TPC will receive single-agent IV chemotherapy, limited to choice of one of the following 7 agents: eribulin, ixabepilone, vinorelbine, gemcitabine, paclitaxel, docetaxel, or nab-paclitaxel.
  Interventions: Drug: Eribulin; Drug: Ixabepilone; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Docetaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: NKTR-102
  Arms: NKTR-102
Drug: Eribulin
  Arms: Treatment of Physician's Choice (TPC)
Drug: Ixabepilone
  Arms: Treatment of Physician's Choice (TPC)
Drug: Vinorelbine
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine
  Arms: Treatment of Physician's Choice (TPC)
Drug: Paclitaxel
  Arms: Treatment of Physician's Choice (TPC)
Drug: Docetaxel
  Arms: Treatment of Physician's Choice (TPC)
Drug: Nab-paclitaxel
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
This is an open-label, randomized, active comparator, multicenter, international Phase 3 study of NKTR-102 versus TPC in patients with metastatic breast cancer who have stable brain metastases and have been previously treated with an anthracycline, a taxane, and capecitabine in either the adjuvant or metastatic setting (prior anthracycline may be omitted if medically appropriate or contraindicated for the patient).

DETAILED DESCRIPTION:
This is an open-label, randomized, active comparator, multicenter, international Phase 3 study of NKTR-102 versus TPC in patients with metastatic breast cancer who have stable brain metastases and have been previously treated with an anthracycline, a taxane, and capecitabine in either the adjuvant or metastatic setting (prior anthracycline may be omitted if medically appropriate or contraindicated for the patient).

In Group A, NKTR-102 will be administered at a dose level of 145 mg/m2 on a q21d schedule as a 90-minute intravenous (IV) infusion on Day 1 of each treatment cycle. In Group B, TPC will be administered per standard of care. Patients randomized to TPC will receive single-agent IV chemotherapy, limited to choice of one of the following 7 agents: eribulin, ixabepilone, vinorelbine, gemcitabine, paclitaxel, docetaxel, or nab-paclitaxel.

This study will randomize approximately 220 patients using a 1:1 randomization ratio and stratification based on geographic region, tumor receptor status, and Eastern Cooperative Oncology Group (ECOG) status. At Screening, the Investigator must determine which TPC will be offered to the patient.

Data will be collected on subsequent anticancer therapies in both treatment groups from the time patients come off the study treatment until the time of primary data analysis for Overall Survival (OS).

An independent data monitoring committee (DMC) will assess interim safety and efficacy data and determine final number of death events needed to provide 80% conditional power based on the zone adaptive design.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, age ≥ 18 years.
* Histologically-confirmed carcinoma of the breast (either the primary or metastatic lesions) for whom single-agent cytotoxic chemotherapy is indicated. Patients may have either measurable or non-measurable disease according to RECIST version 1.1.
* Patients must have a history of brain metastases that are non-progressing.
* For triple-negative breast cancer, a minimum of 1 prior cytotoxic chemotherapy regimen must have been administered for the indication of metastatic disease.Depending on receptor status, 1 or 2 prior cytotoxic regimens are required prior to enrollment in this trial; hormonal and/or human epidermal growth factor receptor 2 (HER2) -targeted agents may be required.
* Have had prior therapy (administered in the neoadjuvant, adjuvant, and/or metastatic setting) with an anthracycline, a taxane, and capecitabine (prior anthracycline can be omitted if not medically appropriate or contraindicated for the patient).
* Last dose of anticancer therapy must have been administered within 6 months of the date of randomization into this study.
* All anticancer- and radiation therapy-related toxicities must be completely resolved or downgraded to Grade 1 or less (neuropathy may be Grade 2 or less).
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Demonstrate adequate organ function obtained within 14 days prior to randomization and analyzed by the central laboratory.
* Women of childbearing potential (WCBP) must agree to use highly effective methods of birth control throughout the duration of the study until 6 months following the last dose of study drug.
* Males with female partners of child-bearing potential must agree to use a barrier contraception (e.g., condom with spermicidal foam/gel/film/cream/suppository) throughout the duration of the study until 6 months following the last dose of study drug; in addition to their female partner using either an intrauterine device or hormonal contraception and continuing until 6 months following the last dose of study drug. Male patients should not donate sperm until 6 months following the last dose of study drug.

Exclusion Criteria:

* Last dose of anticancer therapy (including HER2-targeted therapy) within 14 days prior to randomization.
* High-dose chemotherapy followed by stem cell transplantation (autologous or allogeneic).
* Major surgery within 28 days prior to randomization.
* Concomitant use of any anticancer therapy or use of any investigational agent(s).
* Received prior treatment for cancer with a camptothecin-derived agent.
* Lesions on imaging, by cerebrospinal fluid or with neurological findings that are consistent with leptomeningeal disease or meningeal carcinomatosis.
* Chronic or acute GI disorders resulting in diarrhea of any severity grade.
* Patients who are pregnant or lactating, plan to get pregnant, or have a positive serum pregnancy test prior to randomization.
* Enzyme-inducing anti-epileptic drugs (EIAEDs) within 14 days of randomization.
* Hepatitis B or C, tuberculosis, or HIV.
* Cirrhosis.
* Prior malignancy (other than breast cancer) unless diagnosed and definitively treated more than 5 years prior to randomization.
* Daily use of oxygen supplementation.
* Significant known cardiovascular impairment.
* Prior treatment with NKTR-102.
* Psychiatric illness, social situation, or geographical situation that preclude informed consent or limit compliance.
* Known intolerance or hypersensitivity to any of the products used in this study or their excipients.
* For patients selecting vinorelbine or gemcitabine as the TPC agent, patients may not receive yellow fever vaccine in the 28 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-11; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (19):
  - Investigator Site - Tucson, Tucson, Arizona
  - Investigator Site - Orange, Orange, California
  - Investigator Site - San Francisco, San Francisco, California
  - Investigator Site - Miami, Miami, Florida
  - Investigator Site - Plantation, Plantation, Florida
  - Investigator Site - West Palm Beach, West Palm Beach, Florida
  - Investigator Site - Athens, Athens, Georgia
  - Investigator Site - Baltimore, Baltimore, Maryland
  - Investigator Site - Boston, Boston, Massachusetts
  - Investigator Site - Minneapolis, Minneapolis, Minnesota
  - Investigator Site - Saint Louis, St Louis, Missouri
  - Investigator Site - New York, New York, New York
  - Investigator Site - Chapel Hill, Chapel Hill, North Carolina
  - Investigator Site - Columbus, Columbus, Ohio
  - Investigator Site - Germantown, Germantown, Tennessee
  - Investigator Site - Fort Worth, Fort Worth, Texas
  - Investigator Site - Houston, Houston, Texas
  - Investigator Site - Salt Lake City, Salt Lake City, Utah
  - Investigator Site - Seattle, Seattle, Washington
- Australia (6):
  - Investigatory Site - Albury, Albury, New South Wales
  - Investigator Site - Darlinghurst, Darlinghurst, New South Wales
  - Investigator Site - Wollongong, Wollongong, New South Wales
  - Investigator Site - Subiaco, Subiaco, Western Australia
  - Investigator Site - Box Hill, Box Hill
  - Investigator Site - Nedlands, Nedlands
- Belgium (5):
  - Investigator Site - Brussels, Brussels
  - Investigator Site - Charleroi, Charleroi
  - Investigator Site - Edegem, Edegem
  - Investigator Site - Liege, Liège
  - Investigator Site - Woluwe- Saint-Lambert, Woluwe-Saint-Lambert
- Investigator Site - Montreal, Montreal, Quebec, Canada
- France (6):
  - Investigator Site - Le Mans, Le Mans
  - Investigator Site - Nimes, Nîmes
  - Investigator Site - Paris, Paris
  - Investigator Site - Rennes, Rennes
  - Investigator Site - Rouen, Rouen
  - Investigator Site - Strasbourg, Strasbourg
- Israel (3):
  - Investigator Site - Beersheba, Beersheba
  - Investigator Site - Haifa, Haifa
  - Investigator Site - Tel Aviv, Tel Aviv
- Italy (4):
  - Investigator Site - Milan, Milan
  - Investigator Site - Milano, Milan
  - Investigator Site - Napoli, Napoli
  - Investigator Site - Roma, Roma
- Portugal (2):
  - Investigator Site - Lisboa, Lisbon
  - Investigator Site - Porto, Porto
- Spain (4):
  - Investigator Site - Barcelona, Barcelona
  - Investigator Site - Madrid, Madrid
  - Investigator Site - Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Investigator Site - Sevilla, Seville
- United Kingdom (3):
  - Investigator Site - Bradford, Bradford
  - Investigator Site - Manchester, Manchester
  - Investigator Site - Nottingham, Nottingham

REFERENCES:
- [Derived] Tripathy D, Tolaney SM, Seidman AD, Anders CK, Ibrahim N, Rugo HS, Twelves C, Dieras V, Muller V, Du Y, Currie SL, Hoch U, Tagliaferri M, Hannah AL, Cortes J; ATTAIN Investigators. Treatment With Etirinotecan Pegol for Patients With Metastatic Breast Cancer and Brain Metastases: Final Results From the Phase 3 ATTAIN Randomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):1047-1052. doi: 10.1001/jamaoncol.2022.0514. PMID 35552364
- [Derived] Tripathy D, Tolaney SM, Seidman AD, Anders CK, Ibrahim N, Rugo HS, Twelves C, Dieras V, Muller V, Tagliaferri M, Hannah AL, Cortes J. ATTAIN: Phase III study of etirinotecan pegol versus treatment of physician's choice in patients with metastatic breast cancer and brain metastases. Future Oncol. 2019 Jul;15(19):2211-2225. doi: 10.2217/fon-2019-0180. Epub 2019 May 10. PMID 31074641

RESULTS

PARTICIPANT FLOW:
Groups:
- NKTR-102: NKTR-102 will be administered at a dose level of 145 mg/m2 on a q21d schedule as a 90-minute intravenous (IV) infusion on Day 1 of each treatment cycle.
- Treatment of Physician's Choice (TPC): TPC will be administered per standard of care. Patients randomized to TPC will receive single-agent IV chemotherapy, limited to choice of one of the following 7 agents: eribulin, ixabepilone, vinorelbine, gemcitabine, paclitaxel, docetaxel, or nab-paclitaxel.
Period: Overall Study
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Started | 92 | 86
Completed | 13 | 9
Not Completed | 79 | 77

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC) | Total
Number analyzed (Participants) | 92 | 86 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.13) | 51.9 (10.50) | 53.3 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 86 | 178
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 69 | 60 | 129
  Unknown or Not Reported | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 66 | 57 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 18 | 38
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Grade - ECOG Performance Status
  1. - Fully active, able to carry on all pre-disease performance without restriction
  2. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 25 | 25 | 50
    1 | 67 | 61 | 128
Reproductive Status [Count of Participants; unit: Participants]
  Of Child-Bearing Potential | 16 | 13 | 29
  Surgically Sterile | 11 | 14 | 25
  Post-Menopausal | 65 | 55 | 120
  Other | 0 | 4 | 4
  Missing | 0 | 0 | 0
Pregnancy Test at Screening [Count of Participants; unit: Participants]
  Performed | 29 | 26 | 55
  Positive | 1 | 1 | 2
  Negative | 22 | 24 | 46
  Borderline | 6 | 1 | 7
  Not Performed | 63 | 60 | 123
Height [Mean (Standard Deviation); unit: centimeters] | 162.7 (6.67) | 162.1 (7.73) | 162.4 (7.19)
Weight [Mean (Standard Deviation); unit: kilograms] | 67.16 (17.468) | 65.97 (15.561) | 66.59 (16.539)
Time since Initial Breast Cancer Diagnosis [Mean (Standard Deviation); unit: years] | 8.094 (5.1700) | 6.950 (5.0941) | 7.541 (5.151)
Breast Cancer at Initial Diagnosis [Count of Participants; unit: Participants] — Stage 1: Primary Tumor is less than or equal to 20 mm in greatest dimension
  Stage 2: Primary Tumor is greater than 20 mm but no less than or equal to 50 mm in greatest dimension
  Stage 3: Primary Tumor is greater than 50 mm in greatest dimension
  Stage 4: Tumor of any size with direct extension to the chest wall and/or to the skin (ulceration or skin nodules)
  Participants
    I | 5 | 10 | 15
    II | 41 | 29 | 70
    III | 22 | 17 | 39
    IV | 10 | 16 | 26
    Unknown | 14 | 14 | 28
Cancer Histology at Initial Diagnosis [Count of Participants; unit: Participants]
  Invasive Ductal Carcinoma | 80 | 77 | 157
  Invasive Lobular Carcinoma | 6 | 1 | 7
  Other | 6 | 8 | 14
Estrogen Receptor Status at Initial Diagnosis [Count of Participants; unit: Participants]
  ER Positive | 52 | 49 | 101
  ER Negative | 40 | 34 | 74
  Unknown | 0 | 3 | 3
Progesterone Receptor (PgR) Status at Initial Diagnosis [Count of Participants; unit: Participants]
  PgR Positive | 40 | 42 | 82
  PgR Negative | 50 | 41 | 91
  Unknown | 2 | 3 | 5
Human Epidermal Growth Factor Receptor (HER2) Status at Initial Diagnosis [Count of Participants; unit: Participants]
  HER2 Positive | 15 | 14 | 29
  HER2 Negative | 76 | 66 | 142
  Unknown | 1 | 6 | 7
Estrogen Receptor Status at Last Biopsy [Count of Participants; unit: Participants]
  ER Positive | 47 | 48 | 95
  ER Negative | 38 | 36 | 74
  Unknown | 7 | 2 | 9
Progesterone Receptor Status at Last Biopsy [Count of Participants; unit: Participants]
  PgR Positive | 32 | 31 | 63
  PgR Negative | 51 | 52 | 103
  Unknown | 9 | 3 | 12
HER2 Receptor Status at Last Biopsy [Count of Participants; unit: Participants]
  HER2 Positive | 12 | 13 | 25
  HER2 Negative | 74 | 69 | 143
  Unknown | 6 | 4 | 10
Estrogen Receptor/Progesterone Receptor Status at Last Biopsy [Count of Participants; unit: Participants]
  ER/PgR Positive | 49 | 49 | 98
  ER/PgR Negative | 36 | 35 | 71
  Unknown | 7 | 2 | 9
Time since Initial Brain Metastasis Diagnosis [Mean (Standard Deviation); unit: years] | 1.137 (1.1061) | 1.194 (1.1748) | 1.165 (1.1369)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Patients
Description: To compare Overall Survival (OS) of patients who receive 145 mg/m2 NKTR-102 given once every 21 days (q21d) with OS of patients who receive Treatment of Physician's Choice (TPC). Overall survival is defined as the time from the date of randomization to the date of death from any cause. Patients will be followed until their date of death or until final database closure. Patients who are lost-to-follow-up or are alive at the time of analysis will be censored at the time they were last known to be alive or at the date of event cut-off for OS analysis.
Time Frame: Within 3 years from study start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
months | 7.8 [6.1 to 10.2] | 7.5 [5.8 to 10.4]

2. Secondary Outcome: Progression-Free Survival (Outside the Central Nervous System)
Description: Progression-Free Survival (PFS) is defined as the time from the date of randomization to the earliest evidence of documented Progressive Disease (PD) or of death from any cause. The date of global deterioration or symptomatic deterioration will not be used as the date of PD. The assessment of PFS outside the CNS will utilize RECIST criteria v1.1.
Time Frame: Through study completion, an expected average of 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
months | 2.8 [2.0 to 4.1] | 1.9 [1.9 to 2.1]

3. Secondary Outcome: Progression-Free Survival in Brain Metastasis (PFS-BM)
Description: Progression-Free Survival in Brain Metastasis (PFS-BM) is defined as the time from the date of randomization to the earliest evidence of documented Progressive Disease (PD) per Response Assessment in Neuro-Oncology-Brain Metastases (RANO-BM) in brain metastases or death from any cause. The PD will also be determined by the investigator's assessments. Progressive Disease (PD) is defined as at least a 20% increase in the sum of longest diameters of CNS target lesions, taking as reference the smallest sum on study. This included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, at least 1 lesion had to increase by an absolute value of 5 mm or more to be considered progression.
Time Frame: Through study completion, an expected average of 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
months | 3.9 [2.6 to 4.3] | 3.3 [1.9 to 3.7]

4. Secondary Outcome: Progression-Free Survival (Overall)
Description: Progression-free survival (CNS and peripheral) is defined as the time from the date of randomization to the earliest evidence of documented PD in either the CNS or peripheral (using RANO-BM) or death from any cause. The PD will be determined by both the investigator's and the central imaging facility assessments. The same statistical methods that were used for PFS and PFS-BM will be used for PFS (Overall). Progressive Disease (PD) is defined as at least a 20% increase in the sum of longest diameters of CNS target lesions, taking as reference the smallest sum on study. This included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, at least 1 lesion had to increase by an absolute value of 5 mm or more to be considered progression.
Time Frame: Through study completion, an expected average of 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
months | 2.1 [1.9 to 3.7] | 1.9 [1.8 to 2.0]

5. Secondary Outcome: Objective Response Rates (ORR) of the NKTR-102 Treatment and the Treatment of Physician's Choice (TPC)
Description: RECIST criteria for lesions outside the Central Nervous System (CNS); RANO-BM criteria for CNS lesions) based upon the best response as assessed by the central imaging facility. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR is calculated as the sum of CR and PR. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Through study completion, an expected average of 1 year
Population: 156 patients had measurable disease by RECIST v 1.1 at baseline and were included in the Response Evaluable population for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 83 | 73
Participants
  Objective Response Rate (CR+PR) | 4 | 2
  Stable Disease | 16 | 5
  Progressive Disease | 38 | 32
  Not Evaluable | 18 | 30
  Missing | 7 | 4

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate will be defined as the proportion of patients having a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) for at least 4 months (≥ 120 days). CR is defined as disappearance of all target lesions for at least 4 weeks with no new lesions, not use of corticosteroids, and patient was stable or improved clinically. PR is defined as at least a 30% decrease in the sum of longest diameters sustained for at least 4 weeks, no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: For at least 4 months, with an expected average of 1 year
Measure: Number; unit: participants
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
participants
  # of Patients who achieved Complete Response | 0 | 0
  # of Patients who achieved Partial Response | 6 | 6
  # of Patients who have Stable Disease >= 120 days | 17 | 5
  # of Patients who achieved Clinical Benefit Rate (CBR) | 23 | 11

7. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) outside the CNS will be defined as the time from first documented CR or PR until the earliest evidence of disease progression per RECIST v1.1 or death from any cause. CR is defined as disappearance of all target lesions for at least 4 weeks with no new lesions, not use of corticosteroids, and patient was stable or improved clinically. PR is defined as at least a 30% decrease in the sum of longest diameters sustained for at least 4 weeks, no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Through study completion, an expected average of 1 year
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 83 | 73
months | 7.4 [7.3 to 16.4] | 3.5 [3.5 to 3.5]

8. Secondary Outcome: Compare Health-Related Quality of Life (HRQoL) Using the European Organisation for Treatment of Cancer (EORTC) Quality of Life Core 30 (QLQ-C30) Module With the Brain Neoplasms 20-question (BN-20) Subscale.
Description: The EORTC QLQ-BN20 Scale has a series of 20 questions each of which involve reporting a scale from 1-4. It is an increasing scale where a score of one indicates "not at all" while a score of four indicates "very much". The minimum score is 20 and the maximum score is 80. The higher the score the worse the outcome.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 for NKTR-102 or 28 days for TPC] and end of Cycle 44.
Population: As the trial progressed, some patients discontinued study treatment as a result of progressive disease, non-PD AE, patient decision, or physician decision.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 79 | 63
Units on a Scale
  QLQ-C30 Score at Baseline | 57.59 (21.607) | 52.25 (24.236)
  QLQ-C30 Score at End of Treatment, approximately 1 year: number analyzed (Participants) | 44 | 35
  QLQ-C30 Score at End of Treatment, approximately 1 year | 46.97 (24.582) | 52.38 (24.801)

9. Secondary Outcome: Compare Health-Related Quality of Life (HRQoL) Using the the EuroQoL 5D (EQ-5D-5L™)
Description: The EQ-5D-5L scale is used to measure health by having a patient answer a series of questions. There are a series of 5 questions each of which is scaled from a score of 4-20 in increasing increments of 4. The scale is numbered from 0 to 100 where 100 means the beast health you can imagine and 0 means the worst health.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 80 | 63
Units on a Scale
  EQ-5D-5L Score at Baseline | 61.41 (19.739) | 60.33 (23.004)
  EQ-5D-5L Score at End of Treatment, approximately 1 year: number analyzed (Participants) | 45 | 35
  EQ-5D-5L Score at End of Treatment, approximately 1 year | 56.53 (23.467) | 61.60 (20.858)

10. Secondary Outcome: Compare Health-Related Quality of Life (HRQoL) Using the Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory scale utilizes a series of 4 questions. The first three are scored with a scale from 1-10. The fourth question has 6 six sub components each of which are scored with a scale of 1-10. For every scale, a score of 0 indicates no fatigue/interference where a score of 10 indicates as bad as you can imagine. A patient's score can range from 0 to 100 where 0 indicates the best outcome and 100 indicates the worst.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 79 | 62
Units on a Scale
  BFI Score at Baseline | 4.18 (2.264) | 4.04 (2.401)
  BFI Score at End of Treatment, approximately 1 year: number analyzed (Participants) | 42 | 34
  BFI Score at End of Treatment, approximately 1 year | 4.83 (2.476) | 4.74 (2.373)

11. Secondary Outcome: Magnitude of Clinical Benefit Assessed by ESMO-MCBS Derived From Overall Survival
Description: The magnitude of clinical benefit of NKTR-102 is assessed by the European Society for Medical Oncology Magnitude of Clinical Benefit Scale (ESMO-MCBS) (v1.0). The scale is graded 5, 4, 3, 2, 1, where grades 5 and 4 represent a high level of proven clinical benefit, and grade 1 represents no clinical benefit. To determine the magnitude of clinical benefit when the median OS with the standard of treatment is ≤ 1 year, the score is derived from the Hazard Ratio (HR) of Overall Survival, overall survival gain, and QoL improvement between two treatment arms. Values reported in the data table are Overall Survival values.
Time Frame: Through study completion, within 3 years from study start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 92 | 86
months | 7.8 [6.1 to 10.2] | 7.5 [5.8 to 10.4]
Statistical Analysis 1: Comparison: NKTR-102 vs Treatment of Physician's Choice (TPC); Test type: Other; ESMO-MCBS (v1.0) = 1

12. Secondary Outcome: Number of Participants With Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.3
Description: The number of participants with adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.3
Time Frame: Through study completion, an expected average of 1 year
Population: 167 patients received at least one dose of study treatment and were included in the Safety population for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 90 | 77
Participants | 90 | 76

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over the entire course of the study or approximately 2 years and 8 months.
Description: 167 patients received at least one dose of study treatment and were included in the Safety population.
Arm/Group | NKTR-102 | Treatment of Physician's Choice (TPC)
All-Cause Mortality (participants affected / at risk) | 2/90 | 0/77
Serious Adverse Events (participants affected / at risk) | 33/90 | 24/77
Other Adverse Events (participants affected / at risk) | 90/90 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 (N=90) | Treatment of Physician's Choice (TPC) (N=77)
Colitis Grade 2 (Gastrointestinal disorders) | 1 | 0
Brain Edema Grade 3 (Nervous system disorders) | 1 | 0
Leukopenia Grade 4 (Immune system disorders) | 1 | 0
Neutropenia Grade 4 (Immune system disorders) | 3 | 0
Esophagitis Grade 3 (Gastrointestinal disorders) | 1 | 0
Pneumonia Grade 3 (Infections and infestations) | 1 | 1
Device Related Infection Grade 4 (Infections and infestations) | 1 | 0
Neutropenic Sepsis Grade 3 (Infections and infestations) | 1 | 0
Hyponatremia Grade 3 (Metabolism and nutrition disorders) | 1 | 1
Malaise Grade 3 (Nervous system disorders) | 1 | 0
Atrial Fibrillation Grade 3 (Cardiac disorders) | 1 | 0
Viral Gastroenteritis Grade 3 (Infections and infestations) | 1 | 0
Vomiting Grade 2 (Gastrointestinal disorders) | 3 | 1
Diarrhea Grade 3 (Gastrointestinal disorders) | 5 | 0
Dehydration Grade 3 (Metabolism and nutrition disorders) | 2 | 0
Hip Fracture Grade 3 (Musculoskeletal and connective tissue disorders) | 1 | 2
Urinary Tract Infection Grade 3 (Infections and infestations) | 1 | 1
Intestinal Obstruction Grade 3 (Gastrointestinal disorders) | 1 | 0
Nausea Grade 2 (Gastrointestinal disorders) | 0 | 1
Fatigue Grade 2 (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal Pain Grade 2 (General disorders) | 0 | 1
Dysphagia Grade 3 (General disorders) | 0 | 1
Esophageal Candidiasis Grade 3 (Infections and infestations) | 0 | 1
Bacteremia Grade 4 (Infections and infestations) | 0 | 1
Contusion Grade 3 (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 2
Febrile Neutropenia Grade 3 (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic Anemia Grade 3 (Immune system disorders) | 0 | 1
Cardiac Tamponade Grade 4 (Cardiac disorders) | 0 | 1
Blindness Grade 3 (Eye disorders) | 0 | 1
Colitis Grade 3 (Gastrointestinal disorders) | 3 | 0
Vomiting Grade 3 (Gastrointestinal disorders) | 0 | 1
Neutropenic Colitis Grade 4 (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Grade 3 (General disorders) | 0 | 1
Generalized Physical Health Deterioration Grade 3 (General disorders) | 1 | 0
Generalized Physical Health Deterioration Grade 5 (General disorders) | 1 | 0
Asthenia Grade 3 (General disorders) | 1 | 0
Fatigue Grade 3 (General disorders) | 0 | 1
Bile Duct Stone Grade 3 (Hepatobiliary disorders) | 1 | 0
Cholecystitis Grade 3 (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal Grade 3 (Hepatobiliary disorders) | 1 | 0
Hepatic Failure Grade 3 (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinemia Grade 3 (Hepatobiliary disorders) | 0 | 2
Pneumonia Grade 5 (Infections and infestations) | 1 | 0
Cellulitis Grade 3 (Infections and infestations) | 1 | 0
Device Related Sepsis Grade 4 (Infections and infestations) | 1 | 0
Lung Infection Grade 3 (Infections and infestations) | 1 | 0
Escherichia Sepsis Grade 3 (Infections and infestations) | 0 | 1
Pyoderma Grade 3 (Infections and infestations) | 0 | 1
Fall Grade 3 (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil Count Decrease Grade 4 (Investigations) | 0 | 1
Failure to Thrive Grade 3 (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia Grade 3 (Metabolism and nutrition disorders) | 0 | 1
Groin Pain Grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasm Grade 3 (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture Grade 3 (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain Grade 3 (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness Grade 3 (Nervous system disorders) | 1 | 0
Epilepsy Grade 2 (Nervous system disorders) | 1 | 0
Fine motor skill dysfunction Grade 2 (Nervous system disorders) | 1 | 0
Hypoesthesia Grade 2 (Nervous system disorders) | 1 | 0
Paresthesia Grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure Grade 2 (Nervous system disorders) | 1 | 1
Syncope Grade 3 (Nervous system disorders) | 1 | 0
Status Epilepticus Grade 3 (Nervous system disorders) | 0 | 1
Confusional State Grade 2 (Psychiatric disorders) | 1 | 0
Confusional State Grade 3 (Psychiatric disorders) | 0 | 1
Mental Status Changes Grade 3 (Psychiatric disorders) | 1 | 0
Hallucination Grade 4 (Psychiatric disorders) | 0 | 1
Pleural Effusion Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis Grade 4 (Vascular disorders) | 0 | 1
Influenza Grade 4 (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 (N=90) | Treatment of Physician's Choice (TPC) (N=77)
Nausea (General disorders) | 54 | 31
Diarrhea (Gastrointestinal disorders) | 66 | 15
Vomiting (General disorders) | 34 | 17
Constipation (Gastrointestinal disorders) | 24 | 20
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 19 | 11
Upper Abdominal Pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Stomatitis (Infections and infestations) | 4 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 5
Abdominal Distension (Gastrointestinal disorders) | 7 | 1
Flatulence (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Fatigue (General disorders) | 36 | 26
Asthenia (General disorders) | 28 | 16
Pyrexia (Gastrointestinal disorders) | 6 | 7
Oedema Peripheral (Gastrointestinal disorders) | 6 | 5
Pain (General disorders) | 5 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 33 | 14
Hypokalemia (Metabolism and nutrition disorders) | 16 | 4
Dehydration (Metabolism and nutrition disorders) | 9 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Headache (Nervous system disorders) | 18 | 9
Dizziness (Nervous system disorders) | 9 | 4
Neuropathy Peripheral (Nervous system disorders) | 3 | 9
Dygeusia (Nervous system disorders) | 7 | 2
Seizure (Nervous system disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 17 | 18
Anemia (Blood and lymphatic system disorders) | 11 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 3
Neutrophil Count Decreased (Investigations) | 6 | 10
Aspartate Aminotransferase Increased (Investigations) | 5 | 9
Weight Decreased (Investigations) | 13 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 9
Platelet Count Decresed (Investigations) | 3 | 4
White Blood Cell Count Decreased (Investigations) | 2 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Urinary Tract Infection (Infections and infestations) | 8 | 3
Insomnia (Psychiatric disorders) | 8 | 5
Anxiety (Psychiatric disorders) | 2 | 6
Depression (Psychiatric disorders) | 6 | 2
Vision Blurred (Eye disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02915744/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02915744/SAP_001.pdf